CLINICAL TRIAL: NCT04430946
Title: Comparison of Postpradial Gut Hormone and Metabolic Responses Between Patients With Type 1 Diabetes Mellitus and Healthy Controls
Brief Title: Postprandial Gut Hormone Responses in Patients With Type 1 Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Alexandros Kokkinos, Associate Professor in Internal Medicine, National and Kapodistrian University of Athens
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: GutT1DM
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: type1diabetes; Hunger; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Lean patients with type 1 diabetes (Experimental): Test meal consumed within 10 minutes
  Interventions: Diagnostic Test: Standardized test meal
- Obese patients with type 1 diabetes (Experimental): Test meal consumed within 10 minutes
  Interventions: Diagnostic Test: Standardized test meal
- Lean healthy control subjects (Active Comparator): Test meal consumed within 10 minutes
  Interventions: Diagnostic Test: Standardized test meal
- Obese healthy control subjects (Active Comparator): Test meal consumed within 10 minutes
  Interventions: Diagnostic Test: Standardized test meal

INTERVENTIONS:
Diagnostic Test: Standardized test meal — A test meal of ~700 kcal consisting of protein and fat will be consumed within 10 minutes

SUMMARY:
The study will compare the postprandial responses to a test meal between subjects with type 1 diabetes and healthy control subjects, in terms of gut hormone levels, meal induced thermogenesis, hunger and satiety perception, as well as futher metabolic parameters.

DETAILED DESCRIPTION:
Aim of the study

To compare the acute effect of the consumption of a test meal on satiety, gastrointestinal hormones' response, post-meal thermogenesis, and further metabolic parameters in lean patients with type 1 diabetes mellitus (T1DM), obese patients with T1DM, and healthy lean and obese controls.

Study subjects:

Four groups of participants will be recruited, consisting of 15 lean healthy subjects (BMI <25 kg/m2), 15 obese healthy subjects, 15 lean patients with T1DM (BMI <25 kg/m2), and 15 obese patients with T1DM (BMI ≥ 30kg/m2). Groups will be matched for age and sex. Healthy volunteers will be recruited from the community, and diabetic individuals from our diabetes clinic. Eligibility criteria will include 18-65 years of age, no use of medications affecting appetite and stable weight (no fluctuations exceeding 5 kg the last 3 months.

Methods:

Demographic data and anthropometric measurements will be collected on the day of visit. Fasting blood samples will be collected for measurement of plasma glucose, insulin, triglycerides, GIP, GLP-1, PYY (total), ghrelin (total). VAS for hunger and satiety will be completed in the fasting state. Participants will then consume a test meal of ~700 kcal consisting of protein and fat (no carbohydrates) within 10 minutes. Blood samples will be drawn and VAS scales completed postprandially at 30, 60, 90, 120, 150, 180 min. RMR measurements using indirect calorimetry will be performed in the fasting state, 1 hour and 3 hours postprandially to assess meal induced thermogenesis. Postprandial responses for these parameters will be assessed as area under the curve (AUC).

Patients with T1DM treated with basal- bolus insulin therapy will receive their regular basal insulin dose and patients on an insulin pump will be kept on their basal rate of insulin infusion. In case of fasting hyperglycemia, the session will be canceled.

Postrpandial glucose excursion will be treated with fast acting insulin.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* BMI >30 kg/m2 for the obese groups

Exclusion Criteria:

* Diabetic neuropathy
* Malignancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-08-25 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Gut peptide hormone responses | 3 hours
  Postprandial responses of ghrelin, PYY, GLP-1, Glicentin, Oxyntomodulin measured as area under the curve (AUC)

SECONDARY OUTCOMES:
Meal induced thermogenesis | 3 hours
  Change in basal metabolic rate after meal consumption as assessed by indirect calorimetry

CONTACTS AND LOCATIONS:
Overall Officials: Alexandros Kokkinos, Principal Investigator — First Department of Propaedeutic Medicine, Laiko General Hospital
Locations (1):
- Diabetes Clinical Research Laboratory, 1st Department of Propaedeutic Internal Medicine, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boutari C, Stefanakis K, Simati S, Guatibonza-Garcia V, Valenzuela-Vallejo L, Anastasiou IA, Connelly MA, Kokkinos A, Mantzoros CS. Circulating total and H-specific GDF15 levels are elevated in subjects with MASLD but not in hyperlipidemic but otherwise metabolically healthy subjects with obesity. Cardiovasc Diabetol. 2024 May 18;23(1):174. doi: 10.1186/s12933-024-02264-5. PMID 38762719
- [Derived] Stefanakis K, Kokkinos A, Simati S, Argyrakopoulou G, Konstantinidou SK, Kouvari M, Kumar A, Kalra B, Mantzoros CS. Circulating levels of all proglucagon-derived peptides are differentially regulated postprandially by obesity status and in response to high-fat meals vs. high-carbohydrate meals. Clin Nutr. 2023 Aug;42(8):1369-1378. doi: 10.1016/j.clnu.2023.06.026. Epub 2023 Jun 28. PMID 37418844